CLINICAL TRIAL: NCT06990698
Title: A Phase 1 First-In-Human Study to Investigate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics Activity of FP008 in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study to Investigate FP008 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhuhai Fapon Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP008-CT1001
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FP008 for injection (Experimental)
  Interventions: Drug: FP008 for injection

INTERVENTIONS:
Drug: FP008 for injection — FP008 should be administered intravenous weekly. Six FP008 dose levels are planned to evaluated.

SUMMARY:
The goal of the phase 1 study is to evaluate the safety, efficacy, pharmacokinetics, and pharmacodynamics activity of FP008 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), multicenter, open-label, dose escalation and dose expansion Phase 1 study of FP008 injection in subjects with advanced solid tumors. This study will evaluate the safety, tolerability, PK, PD, immunogenicity, and preliminary antitumor activity of FP008.

The study consists two parts: Part 1 (dose escalation phase) will evaluate the safety, tolerability, PK, PD, immunogenicity, and preliminary antitumor activity of FP008 treatment, and to estimate the DRDE(s) of FP008. Part 2 (Dose expansion phase) will evaluate the safety, tolerability, PK, PD, immunogenicity, and efficacy at the different DRDE(s)/schedule(s) of FP008 in subjects with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written ICF and be able to comply with the protocol.
2. Male and female subjects ≥18 years of age.
3. Life expectancy of >3 months.
4. Laboratory values for sufficient organ function at screening.
5. Toxicity from prior antitumor treatment has resolved to ≤Grade 1 as defined by NCI CTCAE v5.0.
6. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to the start of FP008.
7. Male or women of childbearing potential, if sexually active, must agree to use contraception considered adequate and appropriate by the investigator during the period of study drug administration and for at least 5 months after the last dose of FP008.
8. ECOG performance status of 0 to 1.
9. Histologically or cytologically confirmed malignancy diagnosis and at least one measurable documented advanced/unresectable or metastatic solid tumor as assessed by RECIST v1.1.
10. Documented progressive disease, refractory/resistance/intolerant to standard therapy (documented the reason(s) why they are intolerant to standard therapy by the investigator), or there is no standard therapy.

Exclusion Criteria:

1. Subjects who have received other IL-10 agents.
2. A history of other malignancies other than basal cell carcinoma of skin, squamous cell carcinoma of skin, non-muscle invasive bladder cancer, thyroid papillary carcinoma or carcinoma in situ of the cervix that have been cured for 2 years after effective treatment.
3. Received live vaccine within 30 days prior to the first dose of FP008.
4. Not completely recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of FP008.
5. Known hypersensitivity to either the drug substances or inactive ingredient of FP008.
6. Subjects with diagnosis of immunodeficiency, organ transplant requiring immunosuppressive therapy, or allogeneic bone marrow or hematopoietic stem cell transplant.
7. Daily requirement for corticosteroids within 2 weeks prior to first dose of FP008.
8. Any other medical disorder, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that the investigator considers unsuitable for participation in the study.
9. Cardiovascular dysfunction or clinically significant cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Up to 2 years
Severity (as graded by NCI CTCAE v5.0) of TEAEs leading to discontinuation of study treatment | Up to 2 years
Severity (as graded by NCI CTCAE v5.0) of TRAEs leading to discontinuation of study treatment | Up to 2 years
Severity (as graded by NCI CTCAE v5.0) of SAEs leading to discontinuation of study treatment | Up to 2 years
Severity (as graded by NCI CTCAE v5.0) of irAEs leading to discontinuation of study treatment | Up to 2 years
Severity (as graded by NCI CTCAE v5.0) of AESIs leading to discontinuation of study treatment | Up to 2 years
Severity (as graded by NCI CTCAE v5.0) of AEs leading to discontinuation of study treatment | Up to 2 years

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of FP008 | Up to 2 years
Time to reach maximum plasma concentration (Tmax) of FP008 | Up to 2 years
Area under the curve from time zero to the last measurable time point (AUC0-tlast) of FP008 | Up to 2 years
Area under the curve extrapolated to infinity (AUC0-inf)of FP008 | Up to 2 years
Apparent volume of distribution (V) of FP008 | Up to 2 years
Clearance rate (CL) | Up to 2 years
Maximum plasma concentration during the dosing interval at steady state (Cmax,ss) | Up to 2 years
Minimum plasma concentration during the dosing interval at steady state (Cmin,ss) | Up to 2 years
Terminal elimination half-life (t1/2) of FP008 | Up to 2 years
Incidence of ADA against FP008 | Up to 2 years
Overall response rate (ORR) assessed using RECIST v1.1 and iRECIST | Up to 2 years
Duration of response (DoR) assessed using RECIST v1.1 and iRECIST | Up to 2 years
Disease control rate (DCR) assessed using RECIST v1.1 and iRECIST | Up to 2 years
Progression free survival (PFS) assessed using RECIST v1.1 and iRECIST | Up to 2 years
Time to response (TTR) assessed using RECIST v1.1 and iRECIST | Up to 2 years
Overall survival assessed using RECIST v1.1 and iRECIST | Up to 2 years
Onset time of ADA against FP008. | Up to 2 years
Titer of ADA against FP008. | Up to 2 years
Incidence of Nab against FP008. | Up to 2 years
Onset time of Nab against FP008. | Up to 2 years
Titer of Nab against FP008. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- China (3):
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided